CLINICAL TRIAL: NCT05074147
Title: Three Weeks Versus Six Weeks Antibiotic Therapy for Nonsurgically Treated Diabetic Foot Osteomyelitis : a Multicenter, Randomized, Open-label and Controlled Study
Brief Title: Comparison Between Two Durations of Antibiotherapy for Non-surgically-treated Diabetic Foot Osteomyelitis (CHRONOS-2)
Acronym: CHRONOS-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: logistical and financial problems
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIPH_2019_04
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Osteomyelitis - Foot
Keywords: Diabetes Mellitus; Antibiotic Treatment
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 weeks antibiotherapy (Experimental): Patients are treated 3 weeks with appropriate antibiotics after antibiogram evaluation.
  Interventions: Drug: Reduction in the duration of antibiotic therapy 3 weeks or 6 weeks
- 6 weeks antibiotherapy (Experimental): Patients are treated 6 weeks with appropriate antibiotics after antibiogram evaluation.
  Interventions: Drug: Reduction in the duration of antibiotic therapy 3 weeks or 6 weeks

INTERVENTIONS:
Drug: Reduction in the duration of antibiotic therapy 3 weeks or 6 weeks — Drugs :
  * Rifampin (IP an PO) : 10mg/Kg/12h
  * Ofloxacin (PO) : 200Mg/8h
  * Levofloxacin (PO) : 500mg ot 1g/ twice a day
  * Ciprofloxacin : IV : 400mg/8h if Pseud spp ; 400mg/12h for others Gram-negative bacilli strains; PO : 1gr/12h if Pseud spp ; 750mg/12h for others Gram-negative bacilli strains
  * Clindamycin : 600-900mg/8h
  * Fusidic Acid : 500mg/8h
  * Teicoplanin : 10mg/kg/12h for 5 dosis in combination, then in monotherapy.
  * Ceftasidim : 2g/8h if Pseud spp ; 2g/12h for others Gram-negative bacilli strains
  * Trimethoprim-sulfamethoxazole (800mg/160mg) : once per day if patient < 80Kg ; one and a half per day if patient > 80Kg.
  * Doxycyclin : 200mg/day
  * Minocyclin : 100mg/8h to 12h
  * Ceftriaxon : 1g to 2g/day in IV, IM or SC
  * Cefotaxim : 1g to 2g/day in IV
  * Pristinamycin : 1g thrice a day

SUMMARY:
The aim of this clinical study is to compare the efficacy and tolerance of 3 versus 6 weeks of antibiotherapy in patients with diabetic foot osteomyelitis treated medically.

DETAILED DESCRIPTION:
The fight against multi-drug resistant bacteria is a global matter and a major health public issue. The excessive exposure of microorganisms to drugs increases their ability to develop survival mechanisms, causing an emerging threat and a health challenge.

Several recent studies showed that 18-35% of patients with diabetic foot infections harbored multiply drug-resistance to organisms (MDRO), the most common is Staphylococcus aureus (MRSA). Hospitalization, surgical procedures and long antibiotic therapy induce the development of MDRO or MRSA In diabetic foot, Osteomyelitis (DFO) is a well recognize risk factor for major amputation and mortality rates that occurs in more than 20% of moderate infections and 50% to 60 % of severe infections. In this context, the aim of this study is to evaluated that reducing time of antibiotic administration (3 weeks) is not substantially worse than the current treatment guidelines (6 weeks) in DFO managed nonsurgically.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Informed, written consent obtained from patient
* Patient having the rights to Frenc social insurrance
* For women of childbearing potential : any effective contraceptive is required
* Type 1 or 2 diabetic patients
* Diabetic patients treated non-surgically for an osteomyelitis of the forefoot affecting only one osteoarticular part/radial supported by adequate diagnostic imaging and bone biopsy performed through uninfected tissue.
* Two peripheral pulses or transcutaneous oxygen tension measurement (TcPO2 > 30mmHg) or ankle brachial index (ABI > 0.9)
* Patient without antibiotherapy during 2 weeks before D1.
* Glycated hemoglobin (HbA1C) < 12% ( measured maximum 2 months before D1)
* Use of offloading boot for diabetic foot is feasible

Exclusion Criteria:

* Bone fragmentation, articular destruction requiring bone resection or amputation.
* Gangrene
* More than one osteoarticular part/radial affected
* Contraindication for the use of offloading boot
* Contraindication for bone biopsy
* Contraindication for the full course of antibiotics (allergy or based on RCP)
* Other drug-drug interaction that contraindicated the full course of antibiotics
* Charcot foot
* Patient undergoing radiotherapy of chimiotherapy for malignant neoplasms
* Hepatic insufficiency (ASAT and/or ALAT > 3 times the normal level)
* Any disease or behaviour making impossible to follow the protocol or difficult to interpret the results
* Any disease or context making difficult to allow regular monitoring of the patient
* Participation in other interventional research during the study
* Curator or guardianship of patient placed under judicial protection
* Pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of treated patients achieving remission from the diabetic foot osteomyelitis at the end of follow-up | 12 months
  Remission is defined as one of following events :
  * No relapse of infection at the initial or a contiguous site leading to make a new antibiogram.
  * Absence of pathology exacerbation visible by radiological results (comparison with Day 0)
  * Absence of orthopedic surgery or amputation of the foot infected initially.

SECONDARY OUTCOMES:
Time needed for a complete wound healing in each group. | 12 months
  A wound healing is complete with epithelial wound closure maintained 28 days minimum of the initial site of injury caused by osteomyelitis.
Rates of reinfection at the initial site in each group of patients. | 12 months
  Reinfection is defined by a relapse of infection of soft tissues and osteomyelitis.
Rates of occurrence of a new wound after healing, on the same site initially traited in each group of patients. | 12 months
  A new wound is defined by a skin injury under the malleolus evolving over three weeks.
Rates of occurrence of a new wound after healing on the same foot but not the same infection site in each group of patients. | 12 months
  A new wound is defined by a skin injury under the malleolus evolving over three weeks.
Rates of occurrence of a peripheral neuroathropathy (Charcot foot) in each group of patients. | 12 months
  Neurologic exam includes monofilament test and tuning fork test for assessing the loss of protective sensation.
Rates of amputation in each group of patients. | 12 months
  Minor amputation is defined as an amputation below the ankle (malleolus). Major amputation is defined as an amputation above the ankle (malleolus).
Rates of major amputation in each group of patients. | 12 months
  Major amputation is defined as an amputation above the ankle (malleolus).

CONTACTS AND LOCATIONS:
Overall Officials: Eric M SENNEVILLE, MD, PhD, Principal Investigator — Centre Hospitalier de Tourcoing
Locations (18):
- France (18):
  - Centre Hospitalier de Béthune-Beuvry, Béthune
  - AP-HP Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer
  - Centre Hopitalier Universitaire de Brest, Brest
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier de Compiègne-Noyon, Compiègne
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier de Lens, Lens
  - Centre Hospitalier Universitaire de Lille, Lille
  - GHICL Saint-Vincent de Paul, Lille
  - GHICL Saint-Philibert, Lomme
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - AP-HP Cochin, Paris
  - AP-HP Lariboisière, Paris
  - Centre Hospitalier de Roubaix, Roubaix
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No